CLINICAL TRIAL: NCT06253429
Title: Oxidative Stress in Children and Adolescents With Diabetic Nephropathy and the Role of Adjuvant Alpha-lipoic Acid as an Antioxidant
Brief Title: Alpha-lipoic Acid in Diabetic Nephropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU MS 662/2022
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Thioctic Acid; Tablets; Captopril

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Active Comparator): including pediatric patients with diabetic nephropathy receiving oral alpha-lipoic acid daily.
  The capsule of ALA ( Thiotex 300 mg capsule) contains 300 mg of thioctic acid, manufactured bt Marcyrl Pharmaceutical Industries - Egypt.) The patient will receive 1 capsule twice daily for 3 months. Patients' compliance to therapy will be checked by counting pills.
  oral angiotensin-converting enzyme inhibitors (ACE-Is) captopril 25 mg tablet provided their blood pressure will be maintained within normal range for age
  Interventions: Drug: Thioctic Acid 333 MG Oral Capsule; Drug: Captopril 25Mg Tab
- Control Arm (Placebo Comparator): including pediatric patients with diabetic nephropathy receiving placebo that is similar in appearance to the oral alpha-lipoic acid (Thiotex 300 mg capsule) and oral angiotensin-converting enzyme inhibitors (ACE-Is)(Captopril 25 mg tablet) provided their blood pressure will be maintained within normal range for age
  Interventions: Drug: Captopril 25Mg Tab

INTERVENTIONS:
Drug: Thioctic Acid 333 MG Oral Capsule — Antioxidant compound which serve as a cofactor for mitochondrial respiratory enzymes
  Other Names: Alpha lipoic acid 300 mg tablet
  Arms: Interventional arm
Drug: Captopril 25Mg Tab — Oral angiotensin-converting enzyme inhibitors
  Other Names: Capoten 25 mg tab

SUMMARY:
Endothelial dysfunction in diabetes is a central event in the pathogenesis of different microangioapthic changes. Nephropathy in patients with type 1 diabetes is a severe microvascular complication.

DETAILED DESCRIPTION:
Better understanding of the pathogenesis of microvascular complications in type 1 diabetes have paved the way for novel therapeutic targets and possible adjuvant therapeutic modalities. Oxidative stress is considered a common and important factor that links hyperglycemia with the vascular complications in diabetes, including of diabetic nephropathy (DN).

Alpha lipoic acid (ALA), or thioctacid, is an antioxidant compound which serve as a cofactor for mitochondrial respiratory enzymes. ALA can scavenge free radicals, activate antioxidant systems, and also affect inflammatory markers. It also has unique characteristic. ALA can play as a reduction for oxidized forms of components with antioxidant properties and neutralize reactive oxygen species. Thus, it called as antioxidant of antioxidants

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with type 1 diabetes
* The presence of diabetic nephropathy

Exclusion Criteria:

* Renal impairment due to causes other than diabetes
* Other diabetic complications than nephropathy
* Elevated liver enzymes
* Hypersensitivity to lipoic acid
* Participation in a previous investigational drug study within the 30 days preceding screening

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Total antioxidant capacity and Malondialdehyde | 3 months
  Changes in Total antioxidant capacity and Malondialdehyde
Changes in urinary albumin excretion rate | 3 months
  Changes in urinary albumin excretion rate and HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine I Elhenawy, Principal Investigator — Ain Shams University
Locations (1):
- Pediatrics and Adolescents Diabetes Unit (PADU), Pediatrics Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No